CLINICAL TRIAL: NCT01060709
Title: Does Transcutaneous Carbon Dioxide Partial Pressure (TcCO2) Monitoring Detect Hypoventilation Prior to Current Sedation Monitoring Practices?
Brief Title: Transcutaneous Measurement of Carbon Dioxide Versus Current Sedation Practices in Sedated Patients
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: J.K.Oosterhuis, University Medical Center Groningen,
Other Study IDs: TcCo2-001
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2009-11

CONDITIONS: Colonoscopy
Keywords: Carbon dioxide; TcC02; Hypoventilation; endoscopic; elective colonoscopy and requiring sedation
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- elective colonoscopy and requiring sedation

SUMMARY:
Does transcutaneous carbon dioxide partial pressure (TcCO2) monitoring detect hypoventilation prior to current sedation monitoring practices in order to prevent hypoxemia in sedated patients undergoing colonoscopies?

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring sedation for colonoscopy

Exclusion Criteria:

* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective colonoscopy and requiring sedation
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Does transcutaneous carbon dioxide partial pressure (TcCO2) monitoring detect hypoventilation prior to current sedation monitoring practices in order to prevent hypoxemia in sedated patients undergoing colonoscopies? | one year

SECONDARY OUTCOMES:
To verify if there is an association with the following variables: age, gender, weight, length, ASA-classification, sedation depth (BIS), co-morbidity, diagnostic or therapeutic colonoscopy. | one year

CONTACTS AND LOCATIONS:
Overall Officials: J K Oosterhuis, Drs, Study Director — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands